CLINICAL TRIAL: NCT00557934
Title: Evaluation of Right Ventricular Contractility Reserve Function During Dobutamine Stress in Patients Following Surgical Repair of Tetralogy of Fallot
Brief Title: Right Ventricular Contractility Reserve Following Repair of Tetralogy of Fallot
Acronym: TOF-Cond
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Fördergemeinschaft Deutsche Kinderherzzentren, Bonn, Germany (Unknown)
Responsible Party: Professor Dr. Michael Hofbeck, University Children's Hospital, Tuebingen, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Cond-07-1
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Right Ventricular Dysfunction
Keywords: tetralogy of Fallot; right ventricular dysfunction; pulmonary insufficiency; pulmonary valve replacement; pressure-volume loops; long-term follow-up in tetralogy of Fallot
MeSH Terms: conditions — Ventricular Dysfunction, Right; Tetralogy of Fallot; Respiratory Insufficiency | interventions — Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: dobutamine

INTERVENTIONS:
Other: dobutamine — dobutamine stress (10 µg/kg/min) for 10 minutes during heart catheterization

SUMMARY:
Background: Residual pulmonary regurgitation following repair of tetralogy of Fallot, in particular the use of a transannular patch, has been shown to correlate with the development of right ventricular dysfunction. Optimal timing of pulmonary valve replacement, therefore, is important to preserve right ventricular function. Several recent studies suggested that a threshold of right ventricular end-diastolic volume for intervention, in order to preserve the likelihood of adequate reverse remodeling, is in the region of 150 to 200 ml/m2 body surface area. However, there is evidence that right ventricular function does not always recover following pulmonary valve replacement even if the end-diastolic volume is below this cut-off.

In addition, previous studies suggested that early dysfunction may be present before symptoms occur. However, early dysfunction is difficult to assess.

Methods: Analysis of right ventricular function by pressure-volume loops has been extensively evaluated in experimental studies and is generally considered the optimal way to quantify right ventricular function.

By recording a family of pressure-volume loops during reduction of preload, achieved by temporary balloon occlusion of the inferior caval vein, the contractility can be calculated by the slope of the endsystolic pressure-volume relation (elastance). Changes of contractility following dobutamine infusion could be noted by changes of elastance. The increase of the slope during dobutamine demonstrates the contractility reserve of the right ventricle.

Purpose: To evaluate the right ventricular contractility reserve to determine early ventricular dysfunction after repair of tetralogy of Fallot.

ELIGIBILITY:
Inclusion Criteria:

1. Corrected tetralogy of Fallot or other surgery with involvement of the pulmonary valve, chronic pulmonary regurgitation, dilated right ventricle
2. Patient's age > 4 years
3. Routine cardiac catheterization clinically indicated for deciding therapeutic treatment
4. Informed assent/consent of patients/parent.

Exclusion Criteria:

1. Pregnancy/breast feeding, women of child-bearing age without contraception.
2. Present participation, and/or participation in a clinical study during the last 4 weeks.
3. Illnesses or malfunctions, which exclude a participation in this study after decision of the investigating physician.
4. Other medical, psychological or social circumstances which complicate a regular participation in the study, and/or increase the risk for the patients themselves.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Percentage of change of the maximal elastance (slope of the endsystolic pressure-volume relation)of the right ventricle following dobutamine infusion | 10 minutes after starting dobutamine infusion

SECONDARY OUTCOMES:
Brain natriuretic peptide | at cath study
RV enddiastolic volume index (by MRI) | within the last 6 months before study

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hofbeck, MD, Principal Investigator — University Childrens Hospital, Department of Pediatric Cardiology
Locations (1):
- Department of Pediatric Cardiology, University Childrens Hospital, Tübingen, Baden-Wurttemberg, Germany